CLINICAL TRIAL: NCT03692260
Title: Interfragmentary Gap Following Cannulated Headless Herbert Screw Insertion Using Customized 3-D Surgical Templates Versus Titanium Plate In Reduction & Fixation of Unilateral Minimally Displaced Mandibular Angle Fracture. RCT
Brief Title: Fracture Gap After Herbert Screw Insertion by 3d Stents Vs Titanium Plate(Minimally Displaced Mandibular Angle Fracture)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nevine Alaa Eldine, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-09-29
Record Dates: First submitted 2018-09-27; First posted 2018-10-02 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-09

CONDITIONS: Minimally Displaced Mandibular Angle Fracture

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): 3D stent in Herbert screw insertion vs titanium plate
  Interventions: Procedure: 3D stent in Herbert screw insertion vs titanium plate
- control group (No Intervention): titanium plate

INTERVENTIONS:
Procedure: 3D stent in Herbert screw insertion vs titanium plate — benefit of 3d template in fracture gap
  Arms: intervention group

SUMMARY:
interfragmentary gap measurement using Herbert cannulated headless screw using a 3D surgical customized template versus titanuim plate

DETAILED DESCRIPTION:
* Intervention for each group

  1. Diagnosis

     * for group I and II According to inclusion and exclusion criteria, patients are selected after a comprehensive clinical and radiographic examination and understanding of participant s chief complains.
     * Inspection for the soft tissue laceration, edema, ecchymosis, hemorrhage, cerebrospinal fluid leakage, gingival lacerations, mandible contour deformity, facial asymmetry and the other facial bones bilateral palpation starting from the condylar region descending towards the posterior border of the mandible to look for any tenderness, step deformities or crepitus. Examination of the integrity of the neurosensory and motor function of the injured area.
     * Checking the amount of occlusal discrepancy with complete and comprehensive examination of the dentition.
     * Mandibular movements will also be checked with emphasis on maximal Interincisal opening and midline shift in opening and closing positions.
  2. Surgical planning Group I :participants will be treated using Herbert headless cannulated screw(Zimmer® Herbert™ ,united states of America )Cannulated Bone Screw) using 3d template GroupII :patients are treated using titanium plates (4 or 6 holes according to each case) orthomed ,6th of October,Egypt)
  3. Intra-operative procedures:

     -All of the participants will be treated under general anaesthesia using nasal intubation
     * The occlusion was secured with temporary IMF and the fracture line was exposed and manually reduced.
     * Infiltration Local anesthesia with vasoconstrictor will be injected intraorally at the incision site for hemostatic purposes and pain control.
     * Scrubbing and draping of the patient will be carried out in a standard fashion.
     * An intraoral incision to expose the fracture line. Dissection and reflection to reach the bone For the intervention group planning using the ct software to produce a guiding template of the mandible in the normal position for the insertion of the Herbert screw.

     Reduction of the fracture -Fixation of the fractured segments through Herbert screw using the 3D template fabricated by Plastycad 3diemme Italy(group I), or by using titanium the plate (groupII)

     -Double checking and verification of the occlusion before wound closure.

     -Wounds are debrided and sutured.
  4. Postoperative

     - Cold application at the site of surgery in the form of ice packs 10 minutes every hour in the first 6 hours.

     -Broad spectrum antibiotic therapy in the form of Unasyn 1500 mg vials was given as an IV shot to the patient every 12 hours for 5 days to reduce the risk of infection. (Unasyn®: manufactured by Pfizer, Egypt S.A.E Cairo, A.R.E)
     * Non-steroidal anti-inflammatory drug will be administered in the form of Voltaren 75mg ampoule 3 times daily for 3 days to relief the pain. (Voltaren®: NOVARTIS PHARMA S.A.E. Cairo, under license from: Novartis Pharma AG, Basle, Switzerland.)
  5. Follow up & Evaluation

     Clinical follow up parameters:

     For group I and group II - Dehiscence of the soft tissue and hardware exposure. - Pain over visual analogue scale over first 72 hours.
     * Maximum incisal opening (MIO)
     * Stability of the fractured segments.

     Radiographic follow up parameters:

     - Bone union/nonunion and malunion (OPG).
     * Bone to bone contact via mandible form & border contour (OPG) (3diagnosys 3diemme Italy version 4.2 Any participant that can cause an adverse effect to the intervention/control group will be excluded
     * the patients will receive their panoramic x-ray at the accurate indicated intervals.

     The the MIO will be tested for all patients under the same chair postion using the same caliper, the visual analogue scale to measure the pain will be explained to the patient to prevent any misunderstanding and for the sensory function the patients will be asked to close their eyes before we start to prevent any misleading data as he will not be able to see area we are checking. Those Strategies will be used to improve adherence to intervention protocols.

ELIGIBILITY:
Inclusion Criteria:

* patient age between 20 to 45

  * Patients with minimally displaced angular fracture
  * Patients free from any systemic disease that delay bone healing
  * Patients free from any metabolic bone disease delaying the healing
  * Patients who approved to be included in the trial and signed the informed consent.

Exclusion Criteria:

* .Patients receiving chemotherapy or radiotherapy "due to the risk of low bone quality and healing.(Hopewell, 2003)

  * Patients who refused to be included in the trial

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-25 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
inertfragmentary gap | 3 months as after that time bone remodeling will happen and measuring the interfragmentary gap will be inaccurate
  will be measured using the panoramic xray film on the panoramic radiograph a line was drawn along the fracture and it was divided into 3 equal parts in mm. Perpendicular lines were projected onto the fracture line for reproducible measure points. Measurements of the fracture gap were conducted on these 4 defined points

SECONDARY OUTCOMES:
pain relief | 3 months
  measuring the pain using visual analogue scale (scale fom 0 -10) the patient is asked to pick a number from 0(no pain) till 10(unbearable pain)
nerve sensitivity | 3 months
  nerve sensitivity through neurosensory examination score (score from 1-5) 1means absent to 5 which is intense
maximum incisal opening | 3 months
  using a caliper the measuring unit is in millimeters more opening means better result

CONTACTS AND LOCATIONS:
Overall Officials: Hussein h Abd elrahman, a professor, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
Study results are published as partial fulfillment of the requirements for Phd degree in Oral and maxillofacial surgery by the investigator by cairo university